CLINICAL TRIAL: NCT01079169
Title: Evaluation of the Effect of Cranberry Capsules on the Occurrence of Urinary Tract Infections During Post-acute Rehabilitation of Spinal Cord Injured Patients
Brief Title: Effect of Cranberry Capsules on Urinary Infection Rates in Spinal Cord Injured Patients During Post Acute Rehabilitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated early due to recruitment difficulties
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2009/280
Record Dates: First submitted 2010-02-19; First posted 2010-03-03 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Spinal Cord Injury; Urinary Tract Infection; Rehabilitation
Keywords: urinary tract infection; prevention; rehabilitation; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranberry capsule (Experimental)
  Interventions: Dietary Supplement: Cranberry capsules
- Placebo capsule (Placebo Comparator)
  Interventions: Dietary Supplement: Cranberry capsules

INTERVENTIONS:
Dietary Supplement: Cranberry capsules — Cranberry capsules, 550mg, or placebo capsules, two capsules three times daily during in-patient rehabilitation

SUMMARY:
The purpose of this study is to establish whether cranberry capsules reduce rates of urinary tract infections during initial rehabilitation immediately after spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Previously essentially healthy
2. Newly acquired spinal cord injury, T12 level or higher
3. Receiving in-patient care on the rehabilitation ward.
4. Expected admission duration >= 4 weeks
5. 16 years old or older

Exclusion Criteria:

1. Current or previous disorder that increases the risk of urinary tract infection including diabetes, urological disorder, previous operation on urinary tracts or kidneys, immune dysfunction
2. Severe head injury with impairment of cognitive function
3. Allergy to cranberry
4. Renal failure
5. Warfarin (Coumarin) treatment with unstable INR
6. Current symptomatic urinary tract infection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of symptomatic urinary tract infections per patient per month during in-patient post acute rehabilitation | At end of study

SECONDARY OUTCOMES:
Percentage of in-patient rehabilitation days on which patients were unable to participate in active rehabilitation due to urinary tract infection. | At end of Study
Patient's experience of urinary symptoms in the absence of symptomatic urinary tract infection. | At end of study

CONTACTS AND LOCATIONS:
Overall Officials: Alison K Godbolt, MbChB MD, Principal Investigator — University Hospital Uppsala
Locations (1):
- Dept of Rehabilitation Medicine, University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952